CLINICAL TRIAL: NCT06671795
Title: Improving Intensive Care Through Biobanking: a Strategic Approach to Understanding Post-Intensive Care Syndrome
Brief Title: ICU Biobank: Understanding Post-Intensive Care Syndrome (PICS)
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Akos Tiboldi, Physician, Medical University of Vienna
Other Study IDs: SASICUPICS2012/2023; 101132808 (Other Grant/Funding Number: Innovative Health Initiative Joint Undertaking (IHI JU))
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Post-Intensive Care Syndrome (PICS)
Keywords: Post-Intensive Care Syndrome (PICS); ICU Biobank; Long-term ICU outcomes; Cognitive impairment; Physical impairment; Psychological impairment; Health-related quality of life (HRQoL); Epigenetics in critical care; ICU recovery clinic
MeSH Terms: conditions — postintensive care syndrome; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — The study will retain participant biospecimens, specifically blood samples, and these may be used to extract DNA to explore potential biomarkers related to Post-Intensive Care Syndrome (PICS) and other post-ICU outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore the development and progression of Post-Intensive Care Syndrome (PICS) in adult ICU patients by establishing a biobank of biological samples and outcome data. This biobank-based research is designed to investigate the physical, cognitive, and psychological health outcomes of ICU survivors and their relationship with potential biomarkers. The study population includes adult ICU patients aged 18-65, who have stayed in the ICU for at least 48 hours.

The main questions it aims to answer are:

What is the incidence of PICS and its main components? What risk factors are associated with the development of PICS six months post-ICU discharge? What are the long-term effects of ICU admission on quality of life, cognitive health, and physical function?

Participants will:

Provide blood samples during ICU admission and at follow-up visits at 4-5 weeks, 6 months, and 10-12 months after discharge.

Complete assessments measuring quality of life, cognitive health, anxiety, depression, PTSD symptoms, physical function, and pulmonary function.

Participate in three follow-up visits at the ICU Recovery Clinic after discharge to monitor PICS symptoms and recovery progress.

This study does not involve an intervention but will gather data that could improve our understanding of PICS and inform strategies for post-ICU care. The data collected will be crucial for identifying PICS biomarkers and will contribute to developing targeted, personalized interventions for ICU survivors in the future.

ELIGIBILITY:
Inclusion Criteria:

* ICU stay of at least 48 hours
* Age between 18 and 65 years at the time of ICU admission
* Written informed consent

Exclusion Criteria:

* Transfer from another ICU outside of the Medical University of Vienna
* Patient with a legal guardian
* Homelessness
* Place of residence outside of Austria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 who have been admitted to the Intensive Care Unit (ICU) at the Department of Anesthesia, Intensive Care Medicine, and Pain Medicine at the Medical University of Vienna. Participants are selected based on an ICU stay of at least 48 hours and must provide written informed consent. Patients transferred from other ICUs, those with legal guardians, individuals experiencing homelessness, or those residing outside of Austria are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of PICS and its components | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Incidence of Post-Intensive Care Syndrome (PICS), defined as new or worsened impairments in physical, cognitive, or mental function persisting beyond hospital stay. Patients scoring above/below predefined cut-offs on any of the assessments (detailed below) will be diagnosed with PICS.
Health-related quality of life (HRQoL) using EQ-5D-5L | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  a. The EQ-5D-5L is a responsive, reliable, and robust way of measuring health across a wide range of conditions and populations. It has been translated and validated in 200 languages and includes five dimensions of health: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. The questionnaire will be scored overall and within each category.
Health-Related Quality of Life (HRQoL) using SF-36 | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  HRQoL assessed with SF-36, covering eight health domains. Results will be aggregated into two composite scores: Physical Component Summary (PCS) and Mental Component Summary (MCS), with higher scores indicating a more favorable health state.
Cognitive Function using Montreal Cognitive Assessment (MoCA) | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Cognitive function measured by the MoCA, with scores below 24 indicating impairment. Only patients with prior normal cognitive function are eligible.
Cognitive Function using Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Cognitive decline assessed with IQCODE, a validated informant questionnaire. Scores range from 1 (much improved) to 5 (much worse), with a cutoff average score of ≥3.31 indicating cognitive decline.
Anxiety and Depression Symptoms using HADS | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Anxiety and depression symptoms measured with HADS. Subscale scores ≥8 indicate significant anxiety or depression.
Post-traumatic stress disorder (PTSD) symptoms using Impact of Event Scale-Revised (IES-R) | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  PTSD symptoms measured with the IES-R. Scores range from 0 (not at all) to 4 (extremely), with an average score of ≥1.6 indicating clinically significant PTSD symptoms.
Physical Function using 6-Minute Walk Test (6MWT) | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Deterioration in the 6-Minute Walking Test (6-MWT) defined as a change in the target value of the walking distance calculated using the following equation:
  218 + (5,14 x height - 5,32 x age) - 1,8 x weight + 51,31 x gender (height in cm, age in years, weight in kg, female 0 / male 1)
Physical Function using using Chelsea Critical Care Physical Assessment Tool (CPAx) | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Physical function measured by CPAx, assessing various functional activities (grip strength, respiratory function, moving, sitting, standing, transferring, and stepping). Each domain is scored from 0 to 5, with an overall score from 0 (dependent) to 50 (fully independent).
Pulmonary Function - FEV1/FVC Ratio | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Pulmonary function assessed by FEV1/FVC ratio (Tiffeneau index); a value below the 5th percentile indicates obstructive ventilation disorder.
Pulmonary Function using Total Lung Capacity (TLC) | at 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Pulmonary function assessed by total lung capacity (TLC), where values below the 5th percentile indicate a restrictive ventilation disorder.

SECONDARY OUTCOMES:
Pain and Discomfort using EQ-5D-5L | 4-5 weeks, 6 months and 10-12 months after ICU discharge
  The EQ-5D-5L is a responsive, reliable, and robust way of measuring health across a wide range of conditions and populations. It has been translated and validated in 200 languages and includes five dimensions of health: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. The questionnaire will be scored overall and within each category
Frailty Status using Clinical Frailty Scale | 4-5 weeks, 6 months and 10-12 months after ICU discharge
  Frailty measured by the Clinical Frailty Scale, with scores ranging from 1 (very fit) to 9 (terminally ill). Scores of 1-4 are classified as non-frail; 5-9 as frail.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
The study plans to share de-identified individual participant data (IPD) with other researchers to facilitate additional research on Post-Intensive Care Syndrome (PICS). Shared data will include information related to health outcomes, quality of life assessments, and biomarker findings. Access will be granted through a controlled database managed by the Medical University of Vienna, upon reasonable request and approval by the study's ethics board.
Supporting Information: Study Protocol